CLINICAL TRIAL: NCT04456738
Title: Cascading Dissemination of a Foster Parent Intervention
Acronym: KEEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KEEP60195; R01MH060195 (NIH)
Record Dates: First submitted 2012-02-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Child Welfare; Foster Home Care
Keywords: child behavior; parent training
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent Training (Experimental): 16 weeks of parent training in a group context with 5 to 10 relative and non-relative foster caregivers
  Interventions: Behavioral: Parent Training
- Services as Usual (No Intervention): Foster care services as usual

INTERVENTIONS:
Behavioral: Parent Training — 16 weeks of of parent training led by a trained group facilitator
  Other Names: Parent Management Training
  Arms: Parent Training

SUMMARY:
The primary goal of this study is to test the effectiveness of KEEP (Keeping Foster Parents Supported and Trained), an intervention intended to increase supports and consultation to foster parents, and to evaluate the transferability of the proposed intervention from Oregon to the foster care system in San Diego.

DETAILED DESCRIPTION:
Children in the foster care system are growing in number, are at high risk for psychological problems, and are increasingly challenging to their foster parents. Foster parents who are trying to provide care and nurturing to these children are often doing so without benefit or meaningful or relevant consultation on developmental and mental health issues. The study tests the effectiveness of an intervention intended to increase supports and consultation to foster parents. A major aim of this study was to test the transferability of the proposed intervention from Oregon to the foster care system in San Diego in 3 regions of Health and Human Services. A cascading dissemination model will be employed, where the original developers train and supervise staff in San Diego to implement the intervention, and in the second iteration of the of the intervention, the involvement of the original developers lessened. The intervention is designed to provide foster parents with general support and specific parent management training (PMT), a well-documented and effective intervention approach. In a previous efficacy trial, PMT had positive effects with foster parents in three areas: 1) reduction of child symptoms, 2) lower rates of disruption in foster care (changes in placements for negative reasons), and 3) fewer foster parents in the PMT condition dropped out of providing foster care. Outcomes will be evaluated at multiple levels, including child symptoms, functional behavior, environments, consumer perspectives, and system using a multi-method/multi-agent strategy. Implementation fidelity will be assessed, as will contextual factors, including the organizational climate and social isolation/insularity of the foster parents. It is hypothesized that, compared to controls, foster parents in the intervention group will improve on parenting skills, feel more supported, and have less stress, which in turn will result in more positive child outcomes, including fewer reported child symptoms and higher levels of child functional behavior in three domains (i.e., home, school, with peers). Improvements in foster parent outcomes and child outcomes are both hypothesized to predict system-level outcomes, including child use of mental health services, foster parent retention, and placement disruptions. Contextual factors are expected to impact foster parent outcomes directly and child and system outcomes indirectly, through implementation fidelity.

ELIGIBILITY:
Inclusion Criteria:

* Any child between ages 5 and 12 years in relative or non-relative foster care

Exclusion Criteria:

* Only medically fragile children

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 704 (Actual)
Dates: Start 2000-07; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change in placement disruptions rates for foster placements | 18 months post baseline
  Using child welfare system placement records, rates of disruptions for pre and post time frames are calculated.

SECONDARY OUTCOMES:
Change in child behavior problems as assessed by the Parent Daily Report (PDR) | Baseline, 6 months-, 12 months-, and 18 months post baseline
  The PDR is a brief telephone interview that collects data the number problem behaviors that occurred in the previous 24 hours. This measure is repeated three times at each wave.
Change in rates of reunification with Biological Family as assessed by child welfare system placement records | Baseline through 18 months post baseline
  Using child welfare system placement records, rates of reunification between baseline and 18 months are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Chamberlain, PhD, Principal Investigator — Oregon Social Learning Center
Locations (2):
- United States (2):
  - Child and Adolescent Services Research Center, San Diego, California
  - Oregon Social Learning Center, Eugene, Oregon

REFERENCES:
- [Background] Price JM, Chamberlain P, Landsverk J, Reid JB, Leve LD, Laurent H. Effects of a foster parent training intervention on placement changes of children in foster care. Child Maltreat. 2008 Feb;13(1):64-75. doi: 10.1177/1077559507310612. PMID 18174349
- [Background] Chamberlain P, Price JM, Reid JB, Landsverk J, Fisher PA, Stoolmiller M. Who disrupts from placement in foster and kinship care? Child Abuse Negl. 2006 Apr;30(4):409-24. doi: 10.1016/j.chiabu.2005.11.004. Epub 2006 Apr 5. PMID 16600372
- [Background] Chamberlain P, Price J, Reid J, Landsverk J. Cascading implementation of a foster and kinship parent intervention. Child Welfare. 2008;87(5):27-48. PMID 19402358
- [Background] Chamberlain P, Price J, Leve LD, Laurent H, Landsverk JA, Reid JB. Prevention of behavior problems for children in foster care: outcomes and mediation effects. Prev Sci. 2008 Mar;9(1):17-27. doi: 10.1007/s11121-007-0080-7. Epub 2008 Jan 10. PMID 18185995
- [Background] Degarmo DS, Chamberlain P, Leve LD, Price J. Foster Parent Intervention Engagement Moderating Child Behavior Problems and Placement Disruption. Res Soc Work Pract. 2009 Jul 1;19(4):423-433. doi: 10.1177/1049731508329407. PMID 20072708
- [Result] Price, J., Chamberlain, P., Landsverk, J., & Reid, J. B. (2010). KEEP foster parent training intervention: Model description and effectiveness. Child and Family Social Work, 14, 233-242.